CLINICAL TRIAL: NCT01354652
Title: The Incidence of Lactic Acidosis During Entecavir Treatment in Chronic Hepatitis B Patients With Severe Cirrhosis or Hepatic Failure
Brief Title: Lactic Acidosis During Entecavir(ETV)Treatment
Acronym: ETV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Tenofovir has become available in Korea.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Han Chu Lee, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Hanchu3915
Record Dates: First submitted 2011-05-11; First posted 2011-05-17 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: Lactic Acidosis
Keywords: lactic acidosis; entecavir; lamivudine
MeSH Terms: conditions — Acidosis, Lactic | interventions — entecavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- entecavir (Experimental): Oral 0.5mg/day until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18.
  Participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
  Interventions: Drug: entecavir, lamivudine
- lamivudine (Active Comparator): Oral 100mg/day lamivudine until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18.
  Participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
  Interventions: Drug: entecavir, lamivudine
- no NRTI group (No Intervention): hepatitis C virus associated LC patients for the calculation of lactic acidosis incidence

INTERVENTIONS:
Drug: entecavir, lamivudine — entecavir: 0.5mg/day p.o until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
  lamivudine: 100mg/day p.o until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
  Other Names: Entecavir:baraclude; Lamivudine: zeffix
  Arms: entecavir; lamivudine

SUMMARY:
The purpose of this study is to investigate whether entecavir treatment increases the incidence of lactic acidosis compared to another nucleoside/nucleotide reverse transcriptase inhibitors (NRTI), lamivudine, and/or no NRTI treatment, in patients with cirrhosis or hepatic failure whose Model for End stage Liver Disease (MELD) scores are over 18.

DETAILED DESCRIPTION:
Chronic hepatitis B virus (HBV) infection is the major cause of hepatic failure worldwide. Although the clinical course of HBV infection varies widely, the prognosis of decompensated liver cirrhosis is quite poor and the 5-year survival rate has been estimated to be only 14-35% without treatment. While the ultimate treatment of decompensated cirrhosis is orthotopic liver transplantation (OLT), several studies have suggested that anti-viral therapy can also improve the clinical outcomes in this group of patients.

Entecavir (ETV) is a potent cyclopentyl guanosine nucleoside inhibitor of the HBV polymerase. It has a higher anti-viral potency and a lower resistance rate compared to lamivudine (LAM), telbivudine or adefovir, when used for nucleoside/nucleotide-naïve patients. ETV has been shown to be effective in patients with both hepatitis B envelope antigen (HBeAg)-positive and HBeAg-negative chronic hepatitis B, and compensated liver disease. As for patients with decompensated cirrhosis, the investigators recently reported that ETV can not only induce virological response but also improve underlying hepatic function, and thereby can reduce the need for OLT. The cumulative OLT-free survival at 1 year and 2 years was 87.1% and 83%, respectively with ETV treatment.

Despite this dramatic benefit from ETV treatment, a recent study reported that ETV may induce lactic acidosis in patients with severe hepatic and/or renal function impairment. Lange et al. reported that 5 of 16 patients with severely impaired liver function developed lactic acidosis during ETV treatment. Of note, all the five patients who developed lactic acidosis had MELD scores over 20, and no increased serum lactate concentrations were observed in other 11 patients whose MELD scores were below 18. The Child-Pugh score correlated insufficiently with a risk of lactic acidosis. This result is not contradictory to our previous study, since the investigators did not analyze the incidence of lactic acidosis and the MELD score of the studied patients was relatively low (mean value: 11.5)in our study.

Lactic acidosis has been reported occasionally in association with nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs). NRTIs can induce lactic acidosis via interactions with the mitochondrial DNA polymerase. Until now, most reported cases were human immunodeficiency virus (HIV)-infected subjects treated with several nucleoside inhibitors of the HIV reverse transcriptase. Risk factors include didanosine, stavudine, a combination of the two, female gender, age over 40 years, lower CD4 counts, and shorter duration of therapy (less than 12 months). As for non-HIV-infected cases, there was only one case report of fatal lactic acidosis during combination therapy with adefovir and entecavir prior to the report of Lange et al. Interestingly, in vitro inhibition of mitochondrial DNA polymerase was shown for lamivudine, adefovir and tenofovir, but not for entecavir.

Lactate levels in the blood result from the balance between production and clearance. In normal physiologic conditions, lactate is produced primarily from skeletal muscle, skin, brain, intestine and red blood cells. In severe illness, it can be produced in many other tissues including lung, leukocytes, liver, or intestine. Lactate clearance occurs principally in the liver (60%), kidney (30%), heart and skeletal muscles. For these reasons, though lactic acidosis is typically present in shock states in which oxygen delivery is insufficient to meet cellular demand, elevated blood levels can also result from chronic liver disease and renal impairment. In addition, many other conditions have been reported in association with lactic acidosis even without ongoing evidence of hypoxia or ischemia. Examples are malignancy-related metabolic shifts, systemic inflammatory response, hepatic failure, and various drugs including acetaminophen, NRTIs, metformin, propofol, thiamine deficiency, total parenteral nutrition, and even lactulose. Therefore, in critically ill patients with cirrhosis or hepatic failure, lactic acidosis can result from various causes or in combination, in addition to the NRTIs. First of all, liver failure per se is associated with decreased lactate clearance, which is further aggravated in sepsis or renal failure. The liver can also be a source of lactate production and many medications other than NRTIs can precipitate lactic acidosis. For these reasons, it is not still conclusive whether ETV treatment itself is a direct cause of lactic acidosis in critically ill patients with cirrhosis or hepatic failure, since there was no control group in the study of Lange et al. A similar scenario was observed in a study performed in HIV-infected patients, in which mitochondrial-to-nuclear DNA ratio was compared among non-HIV-infected controls, HIV-infected individuals not on NRTIs, and HIV-infected individuals on NRTIs. In this study, HIV alone affected the mitochondrial-to-nuclear DNA ratio, and therefore resulted in lactic acidosis.

Recently, Wong et al. reported the safety and efficacy of ETV in patients with severe acute exacerbation compared to LAM. In this study, ETV treatment was associated with increased short-term mortality in patients with severe acute exacerbation of chronic hepatitis B but achieved better virological response in the long run. Wong et al. assumed that the cause of increased short-term mortality in ETV-treated patients is due to not only the strong immune response but also lactic acidosis. As such, they suggested that LAM may be initiated first and routine switching to ETV after liver function has improved or the adoption of the roadmap concept are reasonable treatment strategies. However, drug resistance can be a problem in the long term because of the increase of resistance mutation for lamivudine or entecavir later in patients who have the history of exposure to lamivudine before entecavir treatment in the past or have been treated with lamivudine.

Thus, the aim of this study is to investigate whether ETV treatment increases the incidence of lactic acidosis compared to another NRTI, lamivudine, and/or no NRTI treatment, in patients with cirrhosis or hepatic failure whose MELD scores are over 18.

ELIGIBILITY:
1. for ETV or LAM group

   Inclusion criteria:
   * 18 and more than 18 years, and less than 65 years
   * HBV-related liver cirrhosis or acute-on-chronic liver failure
   * Prior documentation of chronic HBV infection at least 6 months before randomization
   * MELD score 18 and more than 18
   * Venous blood lactate level 2 and less than 2 mmol/L

   Exclusion criteria:
   * Age of 65 or older, or younger than 18
   * Patients with acute hepatitis B including acute liver failure
   * Acute-on-chronic liver failure precipitated by acute hepatitis A or acetaminophen intoxication
   * MELD score less than 18
   * entecavir, lamivudine, telbivudine, clevudine, adefovir or tenofovir treatment continued longer than 3 months before entry.
   * Evidence of genotypic or virological resistance to lamivudine, clevudine, telbivudine, or adefovir
   * Patients with elevated venous blood lactate levels more than 2 mmol/L
   * Recent episodes of active infection, hypotension (systolic blood pressure less than 90 mmHg), gastrointestinal or other active bleeding within 2 weeks before entry
   * Any alcohol intake within 2 weeks before entry
   * Recent use of acetaminophen, epinephrine, metformin, iron, isoniazid, propofol, salicylate, sulfasalazine, or valproic acid within 2 weeks before entry. Use of lactulose is permitted.
   * Presence of hepatocellular carcinoma. Patients with hepatocellular carcinoma meeting the Milan criteria can be permitted.
   * Any cancer other than hepatocellular carcinoma except cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated at least 3 years prior to entry is permitted.
   * Patients with HIV infection
   * Female patients in pregnancy
2. for no NRTI group

Inclusion criteria:

* Age of 65 or older, or younger than 18
* Liver cirrhosis or acute-on-chronic liver failure not related with HBV
* MELD score 18 and more than 18
* Venous blood lactate level 2 and less than 2 mmol/L

Exclusion criteria:

* Age of 65 or older, or younger than 18
* Patients with positive HBsAg or IgM anti-HBc
* Acute-on-chronic liver failure precipitated by acute hepatitis A or acetaminophen intoxication
* MELD score less than 18
* Patients with elevated venous blood lactate levels more than 2 mmol/L
* Recent episodes of active infection, hypotension (systolic blood pressure less than 90 mmHg), gastrointestinal or other active bleeding within 2 weeks before entry
* Any alcohol intake within 2 weeks before entry
* Recent use of acetaminophen, epinephrine, metformin, iron, isoniazid, propofol, salicylate, sulfasalazine, or valproic acid within 2 weeks before entry. Use of lactulose is permitted.
* Presence of hepatocellular carcinoma. Patients with hepatocellular carcinoma within Milan criteria can be permitted.
* Any cancer other than hepatocellular carcinoma except cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated at least 3 years prior to entry is permitted.
* Patients with HIV infection
* Female patients in pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han Chu Lee, M.D, Principal Investigator — Department of Internal Medicine, Asan Liver Center, Asan Medical Center, University of Ulsan College of Medicine

RESULTS

PARTICIPANT FLOW:
Groups:
- Entecavir: Oral 0.5mg/day until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18.
  Participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
  entecavir, lamivudine: entecavir: 0.5mg/day p.o until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
  lamivudine: 100mg/day p.o until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
- Lamivudine: Oral 100mg/day lamivudine until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18.
  Participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
  entecavir, lamivudine: entecavir: 0.5mg/day p.o until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
  lamivudine: 100mg/day p.o until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
Period: Overall Study
Arm/Group | Entecavir | Lamivudine | no NRTI Group
Started | 3 | 2 | 0
Completed | 0 | 0 | 0
Not Completed | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entecavir | Lamivudine | no NRTI Group | Total
Number analyzed (Participants) | 3 | 2 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 3 | 2 |  | 5
  >=65 years | 0 | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (6.8) | 38.0 (7.1) |  | 46.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 |  | 1
  Male | 2 | 2 |  | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0
  Not Hispanic or Latino | 3 | 2 |  | 5
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 3 | 2 |  | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 0 | 0 |  | 0
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 3 | 2 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Elevated Venous Lactate Levels More Than 2 mmol/L of Any Etiology
Description: incidence of elevated venous lactate levels more than 2 mmol/L of any etiology until development of lactic acidosis, orthotropic liver transplantation (OLT), death, or improvement of hepatic or renal function to MELD score less than 18 and and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Population: Our study was terminated early with only 5 participant enrolled. We gained lactic acid levels for the 5 patients (all elevated), however we considered that it was not sufficient to be analyzed. Morover, we did not further investigate the etiology for elevated lactic acid levels and secondary etiology-based outcomes are not recorded here.
Measure: Number; unit: participants
Arm/Group | Entecavir | Lamivudine | no NRTI Group
Number analyzed (Participants) | 3 | 2 | 0
participants | 3 | 2 |

2. Secondary Outcome: Incidence of Elevated Venous Lactate Levels More Than 2 mmol/L Directly Related to NRTI
Description: incidence of elevated venous lactate levels more than 2 mmol/L directly related to NRTI until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Population: Secondary outcome assessment was not performed due to early termination of the study.
Groups:
- Lamivudine: Oral 100mg/day lamivudine until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18.
  Participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
  less than 18 and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
  entecavir, lamivudine: entecavir: 0.5mg/day p.o until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score lamivudine: 100mg/day p.o until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
Arm/Group | Entecavir | Lamivudine | no NRTI Group
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Incidence of Elevated Venous Lactate Levels More Than 2 mmol/L Caused by Etiologies Other Than NTRIs
Description: incidence of elevated venous lactate levels more than 2 mmol/L caused by etiologies other than NTRIs until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Population: Secondary outcome assessment was not performed due to early termination of the study.
Arm/Group | Entecavir | Lamivudine | no NRTI Group
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Frequency of Concomitant Prescribed Medications Possibly Associated With Lactic Acidosis Other Than NTRIs
Description: Frequency of concomitant prescribed medications possibly associated with lactic acidosis other than NTRIs until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Population: Secondary outcome assessment was not performed due to early termination of the study.
Arm/Group | Entecavir | Lamivudine | no NRTI Group
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Arterial pH and Anion Gap in Cases With Elevated Blood Lactate Levels (at the Time of Detection and Peak Levels
Description: Arterial pH and anion gap in cases with elevated blood lactate levels (at the time of detection and peak levels until development of lactic acidosis, OLT, death, or improvement of hepatic or renal function to MELD score less than 18 and and participants will be followed for the duration of hospital stay, an expected average of 8 weeks.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Population: Secondary outcome assessment was not performed due to early termination of the study.
Arm/Group | Entecavir | Lamivudine | no NRTI Group
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Overall OLT-free Survival
Description: Overall OLT-free survival until development of OLT and death and participants will be followed for the duration of hospital stay or outpatients visit, an expected average of 12 months
Time Frame: Participants will be followed for the duration of hospital stay or outpatients visit, an expected average of 12 months
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Entecavir | Lamivudine | no NRTI Group
Number analyzed (Participants) | 3 | 2 | 0
day | 411 (311) | 175 (223) |

ADVERSE EVENTS:
Time Frame: at least every week during hospital day upto 2 months
Arm/Group | Entecavir | Lamivudine | no NRTI Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No